CLINICAL TRIAL: NCT01514175
Title: A Pilot Study Comparing the Analgesic Efficacy of IV Ibuprofen and IV Ketorolac
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Culpeper Surgery Center (Other)
Collaborators: Cumberland Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Khalid Athar M.D., Medical Director, Culpeper Surgery Center
Allocation: Not Applicable | Model: Single Group | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KACW1
Record Dates: First submitted 2011-06-14; First posted 2012-01-23 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Pelvic Pain
Keywords: Ketorolac; Caldolor; Chronic Pelvic Pain
MeSH Terms: interventions — Ibuprofen; Ketorolac; Ketorolac Tromethamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- ibuprofen versus ketoralac (Experimental): IV ibuprofen (800 mg intravenous ibuprofen administered intravenously over 10 minutes) will be administered as a single dose prior to surgery at the initiation of anesthesia. A corresponding volume of NS will be administered to the group randomized to ketorolac, at the same time to maintain the study blind.
  Interventions: Drug: IV Ibuprofen; Drug: IV Ketorolac

INTERVENTIONS:
Drug: IV Ibuprofen — Patients will be randomized to receive 800 mg intravenous ibuprofen or 30 mg ketorolac; each of the two treatment groups will consist of 25 patients.
  Other Names: IV Caldolor
Drug: IV Ketorolac — Patients will be randomized to receive 800 mg intravenous ibuprofen or 30 mg ketorolac; each of the two treatment groups will consist of 25 patients.
  Other Names: IV Toradol

SUMMARY:
The primary objective of this study is to compare the efficacy of a single dose of intravenous ibuprofen compared to a single dose of ketorolac for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS).

DETAILED DESCRIPTION:
The primary objective of this study is to compare the efficacy of a single dose of intravenous ibuprofen compared to a single dose of ketorolac for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS).

The secondary objectives of this study are:

* To compare amount of and time to rescue medication in the postoperative period between IV ibuprofen and IV ketorolac treatment groups.
* To compare time to mobility in the postoperative period between IV ibuprofen and IV ketorolac treatment groups.
* To compare time to discharge in the postoperative period between IV ibuprofen and IV ketorolac treatment groups.
* To compare the incidence of adverse events between IV ibuprofen and IV ketorolac treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a preoperative diagnosis which is inclusive of chronic pelvic pain scheduled for Laparoscopic Surgery

Exclusion Criteria:

* Inadequate IV access.
* History of allergy or hypersensitivity to any component of IVIb,ketorolac, aspirin (or aspirin related products), NSAIDs, or COX-2 inhibitors.
* Less than 18 years of age or Greater than 65 years of age.
* Use of analgesics, including NSAIDs, less than 12 hours prior to surgery.
* Patients with active, clinically significant anemia.
* History or evidence of asthma or heart failure.
* Pregnant.
* Inability to understand the requirements of the study, be willing to provide written informed consent (as evidenced by signature on an informed consent document approved by an Institutional Review Board [IRB]), and agree to abide by the study restrictions and to return for the required assessments.
* Refusal to provide written authorization for use and disclosure of protected health information.
* Patients with a history of Chronic Pain Conditions or Syndromes excluding patients with Chronic Pelvic Pain.
* Patients with known OSA

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The efficacy of a single dose of intravenous ibuprofen compared to a single dose of ketorolac for the treatment of postoperative pain as measured by patient pain intensity (Visual Analog Scale, VAS). | One Year

SECONDARY OUTCOMES:
Amount of and time to rescue medication in the postoperative period between IV ibuprofen and IV ketorolac treatment groups | 1 Year
Time to mobility in the postoperative period between IV ibuprofen and IV ketorolac treatment groups | One Year
Time to discharge in the postoperative period between IV ibuprofen and IV ketorolac treatment groups | One Year
Incidence of adverse events between IV ibuprofen and IV ketorolac treatment groups | One Year

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Athar, MD, Principal Investigator — Culpeper Regional Health Systems
Locations (1):
- Culpeper Surgery Center, Culpeper, Virginia, United States